CLINICAL TRIAL: NCT02640625
Title: Adjuvant Mucosal Therapy in HIV-infected Men With Insufficient Response to Antiretroviral Therapy
Brief Title: Improving Prognosis in HIV Infection
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Principal Investigator, Dag Henrik Reikvam, MD PhD, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REK 2015/2125
Record Dates: First submitted 2015-12-16; First posted 2015-12-29 (Estimated); Results first posted 2020-03-27 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-12

CONDITIONS: Human Immunodeficiency Virus
Keywords: HIV; Probiotics; Microbiota; Mucosal immunology; Gut biopsy
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Probiotic compound (Experimental): Lactobacillus rhamnosus GG, Lactobacillus acidophilus, Lactobacillus bulgaricus, Bifidobacterium animalis subsp. lactis, and Streptococcus thermophilus.
  Interventions: Dietary Supplement: Probiotic compound

INTERVENTIONS:
Dietary Supplement: Probiotic compound — Lactobacillus rhamnosus GG, Lactobacillus acidophilus, Lactobacillus bulgaricus, Bifidobacterium animalis subsp. lactis, and Streptococcus thermophilus.

SUMMARY:
The primary objective of this study is to assess the safety of probiotics in cART-treated immunologic non-responder (INR) patients with chronic HIV infection.

The secondary objectives are to i) explore the biological effects of probiotics in combined antiretroviral therapy(cART)-treated INR patient with chronic HIV infection, and ii) investigate differences between cART-treated HIV-infected INR and non-INR patients with regards to gut microbial composition and mucosal barrier function.

ELIGIBILITY:
Inclusion Criteria:

* HIV seropositive >4 years.
* Continuous combined antiretroviral treatment (cART) >4 years.
* Plasma HIV RNA <50 copies/mL >3,5 years.
* Cluster of differentiation(CD)4+ T cell count <400 cells/µL (OR >600 cells/µl) >3.5 years.
* Caucasian
* Signed informed consent and expected cooperation of the patients for the treatment and follow up must be obtained and documented according to International Committee on Harmonization (ICH) Good Clinical Practice (GCP), and national/local regulations.

Exclusion Criteria:

* Plasma hepatitis C (HCV) RNA positive.
* Serum hepatitis B surface antigen (HBsAg) positive.
* Comorbidity of inflammatory bowel disease, coeliac disease or malnutrition.
* Concomitant use of non-steroid anti-inflammatory drugs (NSAID), corticosteroids, disease-modifying antirheumatic drugs, or other anti-inflammatory pharmaceutical substances.
* Concomitant use of antithrombotic pharmaceutical substances
* Regular (weekly) use of any probiotic substance within 3 months prior to inclusion.
* Use of antibiotics within 3 months prior to inclusion.
* Deranged liver function (serum albumin <25 g/L or Child-Pugh ≥10)
* Renal failure (estimated glomerular filtration rate (eGFR) <30 ml/min)
* Heart failure (NYHA class II-IV)
* Intolerance to milk or phenylalanine
* Any reason why, in the opinion of the investigator, the patient should not participate

Ages: 25 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dag Henrik Reikvam, MD PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital (Ullevaal campus), Oslo, Norway

REFERENCES:
- [Derived] Meyer-Myklestad MH, Medhus AW, Stiksrud B, Lorvik KB, Seljeflot I, Hansen SH, Holm K, Hov JR, Kvale D, Dyrhol-Riise AM, Kummen M, Troseid M, Reikvam DH. Probiotics to HIV-Infected Immunological Nonresponders: Altered Mucosal Immunity and Microbial Diversity Restricted to Ileum. J Acquir Immune Defic Syndr. 2022 Jan 1;89(1):77-86. doi: 10.1097/QAI.0000000000002817. PMID 34878437

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Probiotic Compound
Started | 20
Completed | 19
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Groups:
- Probiotic Intervention: HIV positive on cART >4 years with CD4 <400 cells/ml and HIV RNA <50 copies/ml
Arm/Group | Probiotic Intervention
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 1
Age, Continuous [Median (Full Range); unit: years] | 49 [38 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Norway | 20
HBsAg negative AND HCV RNA negative AND no gastrointestinal disorders [Count of Participants; unit: Participants] | 20

OUTCOME MEASURES:

1. Primary Outcome: Adverse Effects
Description: Number of Participants who Experienced Adverse Effects
Time Frame: 10 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Probiotic Intervention
Number analyzed (Participants) | 20
Participants | 1

2. Primary Outcome: Delta HIV Viral Load
Description: Unit og Measure: copies/mL
Time Frame: 8 weeks
Measure: Median (Full Range); unit: copies/mL
Arm/Group | Probiotic Compound
Number analyzed (Participants) | 19
copies/mL | 0 [-2 to 31]

3. Primary Outcome: Delta Blood CD4 Count
Description: Unit of Measure: cells/microL
Time Frame: 8 weeks
Measure: Median (Full Range); unit: cells/microL
Arm/Group | Probiotic Compound
Number analyzed (Participants) | 19
cells/microL | 18 [-372 to 145]

4. Secondary Outcome: Alteration in Gut Microbiota Composition
Description: Explorative (Unit of Measure: Descriptive)
Time Frame: 8 weeks
Reporting Status: Not Posted, anticipated posting 2021-12

5. Secondary Outcome: Alterations in Epithelial Gene Expression
Description: Explorative (Unit of Measure: Descriptive)
Time Frame: 8 weeks
Reporting Status: Not Posted, anticipated posting 2021-12

6. Secondary Outcome: Alterations in Lamina Propria T Cell Subsets
Description: Explorative assays on T cell subsets distribution and function (Unit of Measure: Frequency)
Time Frame: 8 weeks
Reporting Status: Not Posted, anticipated posting 2021-12

7. Secondary Outcome: Alterations in Systemic T Cell Intracellular Signaling
Description: Explorative assays on T cell receptor signaling mechanism (Unit of Measure: Frequency)
Time Frame: 8 weeks
Reporting Status: Not Posted, anticipated posting 2021-12

8. Secondary Outcome: Alterations in Systemic Markers of Immune Activation
Description: Explorative assays on soluble inflammation markers and lymphoid cells activation status (Unit of Measure: Descriptive)
Time Frame: 8 weeks
Reporting Status: Not Posted, anticipated posting 2021-12

ADVERSE EVENTS:
Time Frame: 14 months
Arm/Group | Probiotic Intervention
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 1/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Probiotic Intervention (N=20)
Acute cholecystitis with E. coli bacteremia (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-12-18): https://cdn.clinicaltrials.gov/large-docs/25/NCT02640625/Prot_SAP_000.pdf